CLINICAL TRIAL: NCT01307306
Title: Glucose Control in Severely Burned Patients: Mechanisms and Therapeutic Potential
Brief Title: Glucose Control in Severely Burned Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Marc Jeschke, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ins_met_jeschke
Record Dates: First submitted 2011-01-21; First posted 2011-03-02 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Burns
Keywords: Thermal injury; Chemical Burn; Flame Burn
MeSH Terms: conditions — Burns; Burns, Chemical | interventions — Insulin; Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Insulin (Experimental)
  Interventions: Drug: Humulin R
- Control (No Intervention)

INTERVENTIONS:
Drug: Humulin R — Humulin R (U-100) will be given i.v. The dose given will be adjusted in order to achieve a blood glucose level of 130-140 mg/dl.
  Arms: Insulin
Drug: Metformin — Metformin 850 mg q. 8 hours will be given to decrease blood glucose to 130-140 mg/dl.
  Arms: Metformin

SUMMARY:
The central aim of this application is to determine whether improved outcomes with tight euglycemic control are due to insulin-specific responses. The investigators hypothesize that improving insulin resistance will lead to decreased inflammatory and hypermetabolic responses, as well as restored glucose metabolism, and so result in improved clinical outcome of severely burned patients.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 90 years of age
* >20% TBSA
* Admitted to the burn unit within 120 hours following burn
* At least 1 surgical intervention necessary

Exclusion Criteria:

* death upon admission
* decision not to treat due to burn injury severity
* presence of anoxic brain injury that is not expected to result in complete recovery
* known history of AIDS, ARC, HIV, Hepatitis B-E
* history of cancer within 5 years of malignancy currently under treatment
* inability to obtain informed consent
* previous or existing renal dysfunction, liver disease, or hepatic dysfunction
* pre-existing type I diabetes mellitus
* pregnancy
* allergy to metformin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Perform oral glucose tolerance test | at 1-2 months post-admission, up to 6 months
  Standard fasting oral glucose tolerance test with an intake of 75 g of glucose. Subsequent measurements (in mg/dl) of glucose in blood, insulin and c-peptide will be conducted over 2 hours.
Perform oral glucose tolerance test | assessed at discharge (1-4 months post admission depending on the severity of injury)
  Standard fasting oral glucose tolerance test with an intake of 75 g of glucose. Subsequent measurements (in mg/dl) of glucose in blood, insulin and c-peptide will be conducted over 2 hours.

SECONDARY OUTCOMES:
Measure concentrations of serum cytokines | weekly until discharge (1-4 months post admission depending on severity of injury)
  Inflammatory response will be assessed by measuring the concentrations (in pg/ml)of a panel of serum cytokines (IL-1, IFN, TNF etc.) using the Bio-Plex 17-Plex Suspension assay.
Record the episodes of sepsis | daily until discharge (1-4 months post admission depending on severity of injury)
  Patients will be assessed daily for episodes of sepsis. The total number of episodes over the course of hospital stay will be recorded.
Record the episodes of Pneumonia | daily until discharge (1-4 months post admission depending on severity of injury)
  Pneumonia is defined by new progressive and persistent infiltrate, consolidation or cavitations, inhalation injury based on chest X-ray. We will also follow the guidelines provided by the American Burn Association on the definition of Pneumonia in burn patients. Change in sputum (purulent or increased) will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Jeschke, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Ross Tilley Burn Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada